CLINICAL TRIAL: NCT02940015
Title: Collection of Biological and Environmental Samples and Clinical Data From Anonymous Adult Men and Women for Quality Control and Methods Development and Evaluation (ASCA)
Status: Withdrawn | Type: Observational
Why Stopped: Closed by PI.
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170003; 17-E-0003
Record Dates: First submitted 2016-10-08; First posted 2016-10-20 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Laboratory Assay
Keywords: Quality Control; Urine; Tissue; Normal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anonymous Sample Collection - Adults (ASCA): Healthy Volunteers ages 18 and older

SUMMARY:
Background:

Scientists want to improve new studies on how the environment, diet, and genetic factors affect human health. To do this, they need biological samples and clinical data. They want to find better ways to collect, handle, store, and test these samples and data. This could make them more useful for research.

Objective:

To collect anonymous samples and clinical data from people. To find better ways to collect, handle, store, and test them to support health research.

Eligibility:

Healthy people ages 18 and older

Design:

Participants will complete a screening form by phone or in person. The form could include questions about age, race, ethnicity, menopause status, or pregnancy.

Participants will donate a specific amount of a sample. This could be blood, breast milk, cerumen, ear wax, exhaled breath, hair, mucosal or skin cells, nail clippings, saliva, semen, stool, or urine.

Participants may provide an environmental sample such as dust, water, soil, air, or plant life.

Participants may get kits to collect their samples. They may also donate them at a clinic visit.

Visit will take about 30 minutes. They may include:

Sample collection

Questions about diet, smoking, alcohol use, medication, menstrual cycle, and health

Measurement of body composition, naturally occurring radioactivity, or Doppler blood flow

Moderate exercise

Flexibility, muscle strength, or sensory testing

Participants may be asked to participate several times during the study.

DETAILED DESCRIPTION:
Objective:

We propose a common protocol for use in non-invasive (i.e., minimal risk, not involving general anesthesia or sedation) collection of biological and environmental samples and clinical data from anonymous adult volunteers for methods testing and protocol development, quality control, methods development and evaluation. Individual collections conducted under this protocol will submit actual advertisements, forms and names of persons obtaining consent for IRB expedited review.

Study Population:

This protocol covers recruitment of healthy non-pregnant adults (men and women age 18+) and/or pregnant adult women (age 18+).

Design:

All clinical data and sample collection will be performed by clinical and research professionals as appropriate. Biological samples that may be collected include blood or plasma, breast milk, cerumen, exhaled breath, hair, mucosal and skin cells, nail clippings, saliva, semen, stool and urine. In some cases, lymphocytes will be isolated from blood and immortalized. Clinical data may be collected through non-invasive procedures routinely employed in research and clinical practice, and using medical devices approved for marketing (excluding procedures involving x-rays or microwaves). Clinical data collection may include anthropomorphic measurement, body composition assessment, detection of naturally occurring radioactivity, Doppler blood flow, exhaled breath, flexibility testing, moderate exercise, muscular strength testing, physical sensors, and sensory acuity testing where appropriate given the age, weight and health of the individual. Environmental samples may include dust, water, soil, air, vegetation, and other environmental samples that may be collected without damage to property. Compensation for clinical data and sample donation will depend on the time and effort involved in donation. Samples and clinical data may be collected during a one-time collection, or participants may be asked to provide samples and clinical data on several occasions over a specified period.

Outcome Measures:

The samples and clinical and response data will be used to determine if proposed research designs are feasible and if methods are sufficiently valid and precise to be used in epidemiologic studies. They will also be used for quality control purposes in study sample analysis projects. In epidemiologic studies involving the collection, storage and analysis of laboratory samples, it is essential to evaluate the performance of available assays and to assess the impact of storage and handling on the quality of samples

and laboratory analyses. It is also necessary to determine levels of specific biomarkers in the population to aid in study design as well as willingness of specific population groups to provide necessary samples and data. It is essential 1) to demonstrate that a method is sufficiently reproducible and stable over time such that differences in measurements among individuals in the population can be detected; 2) to evaluate measurement reliability by sending blinded control samples along with study samples to testing laboratories

for quality control purposes; 3) to test proposed laboratories or methods by using replicate samples in order to choose the laboratory or method with the greater precision; and 4) to assess how collection, handling, and storage procedures affect measured levels of specific analytes to allow informed decisions about whether to proceed with a specific analysis; 5) to determine levels and distributions of proposed biomarkers to assess study feasibility and determine appropriate study sample size; and 6) evaluate approaches to recruiting

participants for proposed studies with specific sample collection requirements. Under this protocol, methods may include analyses of genes and gene products, peptides, proteins, lipids, immunologic parameters, hormones, viability of cells, evaporation and dilution effects, chemical toxicants and their metabolites, metals, micronutrients and other analytes.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must be 18 years of age or older and able to provide informed consent. All subjects must be healthy as defined by the American Red Cross - "'Healthy' means that you feel well and can perform normal activities. If you have a chronic condition such as diabetes or high blood pressure, healthy also means that you are being treated and the condition is under control."

EXCLUSION CRITERIA:

No children, fetuses, cognitively impaired persons, or prisoners will be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This protocol covers recruitment of healthy non-pregnant adults (men and women age 18+) and/or pregnant adult women (age 18+).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
The samples and clinical data will be used to ascertain whether data and sample collection, processing techniques, and testing methods are sufficiently valid and precise to be used in specific epidemiologic studies. | will vary by sub study effort
  Evaluations of the performance of available assays; assessments of theimpact of storage and handling on the quality of samples and laboratory analyses; determinations of the levels of specific biomarkers in the population to aid in study design as well as willingness of specific population groups to provide necessary samples and data

CONTACTS AND LOCATIONS:
Overall Officials: Paula S Juras, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)